CLINICAL TRIAL: NCT04118751
Title: Impact of Premature Childbirth on Parental Outcomes During Baby's NICU Stay and Beyond: "Preterm Parents" Study on Polish Cohort
Brief Title: Impact of Premature Childbirth on Parental Outcomes During Baby's NICU Stay and Beyond
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Gdansk (Other)
Responsible Party: Principal Investigator, Łucja Bieleninik, Assistant Professor, University of Gdansk
Other Study IDs: 9/2019
Record Dates: First submitted 2019-10-04; First posted 2019-10-08 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Premature Birth
Keywords: Parental outcomes; Bonding; NICU
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- parents of preterm babies (born before 37 weeks of pregnancy
- parents of full-term babies (over 37 weeks of pregnancy)

SUMMARY:
The main objective of this project is examining whether there is a relationship between preterm delivery and parental' problematic emotional bond in the early postpartum period.

The secondary outcomes are as follows:

* To evaluate whether there are any differences and similarities between fathers' and mothers' level of parental bonding, stress, anxiety, and depression symptoms in case of premature birth.
* To evaluate whether there is a relationship between preterm delivery and the persistence of maternal' problematic emotional bond three months after childbirth.
* To indicate what kind of predictors might affect the parental' problematic bond in the early postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children born below the 37th week of pregnancy (clinical group) or above the 37th week of pregnancy (control group) hospitalised in a neonatal setting during recruitment period
* Which agreed participating to the study after having complete information about it and sign a consent.

Exclusion Criteria:

* Parents may not participate in the study if one of them suffers from a serious mental illness.

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: The investigators will approach parents of preterm babies (born before 37 weeks of pregnancy) and parents of babies born on time (over 37 weeks of pregnancy). Patients will be recruited for the study after delivery and will be enrolled after giving their written consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Bonding between primary caregiver and infant | From date of admitted to a NICU until discharge from hospital, assessed up to 7 days after delivery
  Mean score of both parents of preterm babies hospitalized in NICU and parent of full-term babies on Postpartum Bonding Questionnaire (PBQ). Total score of the PBQ, a parent-rated screening instrument for disorders of the early parent-infant relationship consisting of 25 statements on a six-point Likert scale (each 0-5; sum score ranging from 0 to 125; high = problematic).

SECONDARY OUTCOMES:
Parental depression | From date of admitted to a NICU until discharge from hospital, assessed up to 7 days after delivery
  Mean score of parents of preterm infants hospitalized in NICU on Edinburgh Postnatal Depression Scale (EPDS). The EPDS is a 10-item validated self-report instrument assessing mothers' postpartum depressive symptoms, excluding somatic symptoms of depression that are common in new mothers (such as loss of energy, feeling tired, changes in appetite and sexual drive). Sum scores can range from 0 to 30, with high scores indicating more depressive symptoms.
Parental anxiety | From date of admitted to a NICU until discharge from hospital, assessed up to 7 days after delivery
  Mean score of both parents of preterm infants hospitalized in NICU on Generalized Anxiety Disorder Assessment (GAD-7). The GAD-7 is a self-report 7-item questionnaire serving as a screening tool and severity measure for generalized anxiety disorder. Sum scores can range from 0 to 21, with higher scores indicating higher anxiety.
Parental stress | From date of admitted to a NICU until discharge from hospital, assessed up to 7 days after delivery
  Mean score of both parents of preterm infants hospitalized in NICU on Parental Stress Scale (PSS). PSS is a self-report 18-item questionnaire that assesses stress associated with parenting. Sum scores can range from 18 to 90, with higher scores indicating higher stress.
Bonding between mother and infant | Through study completion, an average of 3 months
  Mean score of both parents of preterm babies hospitalized in NICU and parent of full-term babies on Postpartum Bonding Questionnaire (PBQ). Total score of the PBQ, a parent-rated screening instrument for disorders of the early parent-infant relationship consisting of 25 statements on a six-point Likert scale (each 0-5; sum score ranging from 0 to 125; high = problematic).

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Gdańsk, Gdansk, Poland

REFERENCES:
- [Derived] Bieleninik L, Lutkiewicz K, Jurek P, Bidzan M. Paternal Postpartum Bonding and Its Predictors in the Early Postpartum Period: Cross-Sectional Study in a Polish Cohort. Front Psychol. 2021 Apr 9;12:628650. doi: 10.3389/fpsyg.2021.628650. eCollection 2021. PMID 33897536